CLINICAL TRIAL: NCT07371286
Title: Administration of Fiber as a Dietary Supplement to Improve the Management of Alcohol Withdrawal - Randomized Controlled Open-label Study - FIB-ALC
Brief Title: Administration of Fiber as a Dietary Supplement to Improve the Management of Alcohol Withdrawal
Acronym: FIB-ALC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-A00575-44/1
Record Dates: First submitted 2025-11-24; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder; Supplementation; Intestinal Permeability
Keywords: Alcohol; Dietary fibers; Food supplementation; Intestinal permeability; Misuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm taking food bite-sized pieces containing 16 g of dietary fiber (pectin and inulin) (Experimental): group receiving 16 fiber-enriched bite-sized pieces (16 g of fiber in total: 8 g of pectin and 8 g of inulin)
  Interventions: Dietary Supplement: Administration of fibers as a dietary supplement
- Control arm that will not consume the bite-sized pieces (No Intervention): Patients in this arm will not consume the bite-sized pieces and will follow the usual care protocol

INTERVENTIONS:
Dietary Supplement: Administration of fibers as a dietary supplement — Food bite-sized pieces containing 16 g of dietary fiber (pectin and inulin).
  Arms: Experimental arm taking food bite-sized pieces containing 16 g of dietary fiber (pectin and inulin)

SUMMARY:
The goal of this clinical trial is to demonstrate that a fiber-enriched diet (with a high proportion of inulin and pectin) combined with standard care can reduce intestinal permeability in patients with alcohol use disorder (AUD) aged between 19 and 65.

The hypothesis of our study is that a diet rich in different dietary fibers (mainly inulin and pectin), by modifying the gut microbiota and its metabolites, will induce a decrease in intestinal permeability, restore the composition of the gut microbiota and its metabolites, and further improve abstinence, levels of craving and anxiety, inflammation, steatosis, and hepatic fibrosis in patients with alcohol use disorder.

The study consists of two parallel groups (a group eating fiber-rich snacks every day for 28 days (in addition to their usual care) versus a group not eating any snacks).

Participants will be required to provide stool, blood, and saliva samples, and complete questionnaires.

DETAILED DESCRIPTION:
Our study proposes testing a new therapeutic target for alcohol addiction: the gut microbiota, which could have a major impact on the prognosis for these patients, or for other addictive behaviors. Dietary fiber can modify alcohol-related intestinal dysbiosis and improve alcohol-induced changes in the intestinal barrier. Given the potential life-threatening nature of alcohol dependence, our study is the first to evaluate the effectiveness of a high-fiber diet in reducing alcohol consumption, increasing alcohol abstinence rates, and improving addictive behavior, cravings, and anxiety and depression symptoms in patients with severe alcohol addiction. The secondary objectives will allow us to study certain mechanisms involved in these effects, with a particular focus on the gut-brain axis. Given the difficulty of managing this chronic condition, if our results are positive, dietary fiber and dietary modulation could become an additional therapeutic option for alcohol withdrawal, improving prognosis and directly benefiting these patients. Furthermore, compared to other treatments used for alcohol addiction, fiber, through its mode of action, could also improve alcohol-related complications.

Although there is no official maximum intake for dietary fiber, excessive consumption, especially when the amount is increased dramatically over a short period of time, can cause minor, non-severe side effects such as gas and bloating. However, our intervention will not exceed the maximum recommended fiber intake recommended by scientific societies, which will reduce the risk of adverse effects. The constraints for patients are minimal and mainly involve eating the bite-sized pieces in addition to their usual meals and completing specific questionnaires to determine their impact on diet, addictive behaviors, and quality of life.

Subjects participating in the study will receive fiber-enriched food bite-sized pieces (16 bite-sized pieces/day for a total of 16 g of fiber: 8 g of inulin and 8 g of pectin) developed by Carembouche every day for 28 days. To increase compliance, different flavors will be offered (citrus, coffee, vanilla, chocolate) for the patient to choose from at the time of inclusion. The bite-sized pieces will be packaged in batches, one package per day, to be stored at room temperature. The bite-sized pieces will be supplied by Carembouche and stored in the department in a closed cupboard, away from light and in accordance with the manufacturer's instructions. Patients will receive the bite-sized pieces during their hospital stay and will return home with the quantity needed for the following 7 days. During the visit on day 14, patients will receive the quantity needed for the remaining 14 days of the protocol. The treatment includes a phase of gradual dose increase with 4 bite-sized pieces on day 1, 8 on day 2, 12 on day 3, and 16 from day 4 until the end of the study. During this adaptation period, patients will be able to choose flavors according to their taste preferences.

ELIGIBILITY:
Inclusion Criteria:

* Women or men,
* aged >18 and ≤ 65,
* French-speaking,
* active alcohol users (as defined by the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, DSM-5)
* who agree to be hospitalized for alcohol withdrawal for a period of 7 days
* Affiliated with or eligible for social security.
* Negative pregnancy test (for patients of childbearing age)

Exclusion Criteria:

* any other addictive disorder (except tobacco),
* inflammatory bowel disease or any other chronic inflammatory disease,
* current cancer,
* metabolic diseases such as obesity (BMI ≥ 30 kg/m²) kg/m2) or a history of bariatric surgery,
* severe cognitive impairment (MMSE < 24),
* psychiatric comorbidities including suicide risk,
* cirrhosis or significant fibrosis (≥F2) defined by a Fibroscan value >7.6 kPa,
* pregnancy or breastfeeding,
* taking antibiotics, probiotics, or prebiotics in the 2 months prior to inclusion,
* taking non-steroidal anti-inflammatory drugs or glucocorticoids in the month prior to inclusion.
* taking baclofen, disulfiram, naltrexone, or acamprosate.
* Participation in another interventional study involving human subjects or being in the exclusion period following a previous study involving human subjects, if applicable
* Patients under AME
* Patients under guardianship, trusteeship, or any other legal protection measure

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
50% reduction in plasma levels of circulating sCD14 (a surrogate marker of intestinal permeability and bacterial translocation), measured by enzyme-linked immunosorbent assay (ELISA). | From day 0 to day 28

SECONDARY OUTCOMES:
Markers of intestinal integrity (intestinal permeability and bacterial translocation) assessed by plasma measurements of lipopolysaccharide (LPS). | From day 0 to day 28
Markers of intestinal integrity (intestinal permeability and bacterial translocation) assessed by plasma measurements of lipopolysaccharide binding protein (LPB) | From day 0 to day 28
Markers of intestinal integrity (intestinal permeability and bacterial translocation) assessed by plasma measurements of flagellin. | From day 0 to day 28
Markers of intestinal integrity (intestinal permeability and bacterial translocation) assessed by plasma measurements of faecal albumin. | From day 0 to day 28
Markers of intestinal integrity (intestinal permeability and bacterial translocation) assessed by plasma measurements of zonulin. | From day 0 to day 28
Markers of macrophage and neutrophil activation assessed by plasma assays of sCD163. | From day 0 to day 28
Markers of macrophage and neutrophil activation assessed by plasma assays of sCD206. | From day 0 to day 28
Markers of macrophage and neutrophil activation assessed by plasma assays of HMGB1. | From day 0 to day 28
Markers of macrophage and neutrophil activation assessed by plasma assays of osteopontin. | From day 0 to day 28
Evolution of the microbiome profile using 16s DNA sequencing | From day 0 to day 28
Plasma levels of pro-inflammatory cytokines | From day 0 to day 28
  (CRP, ferritin, transferrin, TNF-α, IL-1β, IL-6, IL-8)
Changes in biological and behavioural markers of alcohol consumption measured by plasma levels of carbohydrate-deficient transferrin (CDT) | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by plasma levels of gamma glutamyltransferase (GGT). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by plasma levels of mean corpuscular volume (MCV). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by the abstinence rate assessed using the Alcohol Timeline Followback (TLFB) method. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in craving intensity assessed by the OCDS (Obsessive-Compulsive Drinking Scale) craving score. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in anxiety intensity as assessed by the Hamilton Anxiety Rating Scale (HARS). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in impulsivity assessed using the Urgency Premeditation Perseverance Sensation (UPPS) impulsive behaviour scale. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in the amount of alcohol consumed as assessed by the TLFB method. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in biological markers of liver function (transaminases, alkaline phosphatase, bilirubin). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by progression of liver fibrosis and steatosis using non-invasive tests, assessed by liver elasticity. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by progression of liver fibrosis and steatosis using non-invasive tests, assessed by controlled attenuation parameter (CAP). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by progression of liver fibrosis and steatosis using non-invasive tests, assessed by biological fibrosis score. | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by quality of life assessed by the 9-point Alcohol Dependence Quality of Life Scale (AlQoL9). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by changes in dietary behaviour assessed by the Food Frequency Questionnaire (FFQ). | From day 0 to day 28
Changes in biological and behavioural markers of alcohol consumption measured by the collection of daily tolerance of adverse effects at each visit. | From day 0 to day 35
  Gastrointestinal symptoms will be measured using a French version of a self-reported questionnaire initially developed by gastroenterologists to assess symptoms of irritable bowel syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Carine PARE, Study Director — Assistance Publique - Hôpitaux de Paris